CLINICAL TRIAL: NCT02002416
Title: Prognostic Value and Clinical Pathology of c-MET Expression and Amplification in Gastric Carcinoma: the Comparison Between the Primary and Metastatic Lesions, Early Stage and Advanced Stage
Brief Title: Prognostic Value and Clinical Pathology of c-MET Expression and Amplification in Gastric Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Vice president, Sun Yat-sen University
Other Study IDs: C-met in gastric cancer; Amgen (Other Grant/Funding Number: Amgen)
Record Dates: First submitted 2013-11-20; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Gastric Cancer
Keywords: C-met expression, gastric cancer, overall survival
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Paraffin-embedded tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metastatic gastric cancer patients: Selecte 100 cases of eligible metastatic gastric cancer patients with primary and metastatic lesion (1:1). Use the immunohistochemistry (IHC) and Fluorescence in situ hybridization (FISH) to detect the status of C-met.
- Early stage gastric cancer: Selected 100 cases of eligible gastric cancer patients with previously early stage gastric cancer

SUMMARY:
The MET oncogene encodes the receptor tyrosine kinase (RTK) for hepatocyte growth factor (HGF) and controls genetic programs leading to cell growth, invasion and protec¬tion from apoptosis. Although the definitive role of MET oncogene is yet to be determined in carcinogenesis of gastric cancer, overexpression and amplification of c-Met has been demonstrated in gastric cancer cell lines. In addition, approximately 10-20% of gastric cancer tissues and up to 40% of the scirrhous histological subtype were shown to harbor increased MET gene copy numbers. Importantly, PHA-665,752, a selective c-Met kinase inhibitor showed significant reduction of established tumor mass in mouse xenografts with GTL16, a gastric cancer cell line with >10-fold MET amplification. Another pivotal study showed that gastric cancer cells with MET amplification were extremely sensitive to PHA-665,752 and implicated a potential role of c-Met protein in developing theranostics in gastric cancer. More and more data indicated that c-Met was an important prognostic factor in gastric cancer.

Gastric cancer is a heterogeneous disease. Does the expression and amplification of c-Met in the primary lesion differ from the metastatic disease? Does the expression and amplification of c-Met in the early disease differ from advanced disease? Till now there is no related report.

Purposes:

* Compare the expression and amplification of c-Met between primary lesion and metastatic lesion together with clinical characteristic, to explore the relationship of c-Met expression and metastatic pattern
* Compare the expression and amplification of c-Met between early stage and metastatic stage, and to explore the role of c-MET in the development of carcinoma

DETAILED DESCRIPTION:
We retrospectively collect the metastatic gastric cancer patients who received a surgical resection of both primary diseases and metastatic lesions during January 2006 and December 2012. Patients are collected based on the following criteria: (1) pathology proven advanced gastric adenocarcinoma; (2) the paraffin-embedded tissues of the primary and metastatic lesions were available (3) full information of follow-up. There are 100 patients suitable for the analysis. c-MET protein expression and amplification are assessed in paraffin-embedded tissues of the primary and metastatic diseases obtained from 100 patients by immunohistochemistry (IHC) and Fluorescence in situ hybridization (FISH). The clinical pathologic data of the patients are also collected for analysis, including: gender, age, Karnofsky performance score (KPS), chemotherapy regimens, tumor locations, Lauren classification, histology subtypes, metastatic sites.

In order compare c-Met expression and amplification between early and advanced stage, we will match 100 early stage (stage I and stage II) patients based on the following criteria (1) pathology proven gastric adenocarcinoma with radical resection; (2) the paraffin-embedded tissues of the primary lesions is available (3) full information of follow-up MET IHC will employ the Dako MET IHC assay and supplied assay protocol and pathology scoring guideline.

MET FISH will also employ the Dako MET FISH assay supplied assay protocol and pathology scoring guideline.

ELIGIBILITY:
Inclusion Criteria:

1. For metastatic gastric cancer patients (1) pathology proven advanced gastric adenocarcinoma; (2) the paraffin-embedded tissues of the primary and metastatic lesions were available; (3) full information of follow-up
2. For early stage gastric cancer patients (1) pathology proven gastric adenocarcinoma with radical resection; (2) the paraffin-embedded tissues of the primary lesions is available; (3) full information of follow-up

Exclusion Criteria:

1. Older than 70 years old or younger than 18 years old
2. without paraffin-embedded tissue
3. without information of follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively collect the metastatic gastric cancer patients who received a surgical resection of both primary diseases and metastatic lesions during January 2006 and December 2012. c-MET protein expression and amplification are assessed in paraffin-embedded tissues of the primary and metastatic diseases obtained from 100 patients by immunohistochemistry (IHC) and Fluorescence in situ hybridization (FISH). In order to compare c-Met expression and amplification between early and advanced stage, we will match 100 early stage (stage I and stage II) patients. MET IHC will employ the Dako MET IHC assay and supplied assay protocol and pathology scoring guideline.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  From the diagnosis to the time of last follow up or death

SECONDARY OUTCOMES:
Positive rate of C-met | 8%
  The positive rate of c-met in the primary and metastastic diseases and in different stage diseases patients

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China